CLINICAL TRIAL: NCT02123537
Title: Functional Electrical Stimulation to Treat Foot Drop in People With Multiple Sclerosis
Brief Title: Treating Foot Drop in People With Multiple Sclerosis Using Electrical Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Riverview Health Centre Foundation (Other)
Responsible Party: Principal Investigator, Dr. Karen Ethans, Director, Spinal Cord Rehabilitation Program, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSFD2014
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Sclerosis; Foot Drop
Keywords: Bioness L300 Foot Drop System; Functional electrical stimulation
MeSH Terms: conditions — Multiple Sclerosis; Peroneal Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bioness L300 Foot Drop System (Experimental): Participants will use the Bioness L300 Foot Drop System for walking daily during the 12 weeks of the study.
  Interventions: Device: Bioness L300 Foot Drop System

INTERVENTIONS:
Device: Bioness L300 Foot Drop System — Participants will use the Bioness L300 Foot Drop System during waking hours for 12 weeks.

SUMMARY:
People with multiple sclerosis (MS) often suffer from foot drop, which impairs their walking ability. Foot drop is the inability to lift the foot during the swing phase of walking. The purpose of this study is to find out if electrical stimulation of the leg, using the Bioness L300 Foot Drop System, can be used to treat foot drop in people with MS. It is expected that using this system will reduce foot drop, and therefore improve walking ability, particularly in the areas of speed, strength, balance and falls.

DETAILED DESCRIPTION:
Due to damage of their central nervous system, people with multiple sclerosis (MS) often develop abnormal gait. One common problem is the inability to lift the foot during the swing phase; this is called foot drop, and is caused by loss of ankle dorsiflexor strength and spasticity of the ankle plantarflexors. Foot drop leads to imbalance and increased risk of falling, due to the foot dragging on the ground. Treating foot drop can result in improved gait, faster walking speeds, improved balance and reduced risk of falling.

Functional electrical stimulation (FES) stimulates either the superficial or deep branches of the common peroneal nerve. This stimulation leads to contraction of the ankle dorsiflexors and evertors, which causes dorsiflexion and eversion of the foot, resulting in the stepping motion of lifting the toes toward the shin. This reduces foot drop, allowing the user to regain a more natural stepping pattern; it also reduces spasticity, strengthens muscles and increases joint range of motion.

The Bioness L300 Foot Drop System consists of three components: a leg cuff worn just below the knee, which provides electrical stimulation to the common peroneal nerve; a gait sensor attached to the shoe, which detects which stage of the gait cycle the foot is in; and a control unit, which is used to adjust the level of stimulation received. These three components communicate wirelessly with each other, so that the electrical stimulation is applied at the appropriate time during each gait cycle.

The study physician will set up the system to optimize stimulation according to each participant's gait and needs, and participants will use the system for 12 weeks. There will be an initial four week adaptation period for using the system. During this first four weeks participants will gradually increase their use of the system until they are using it all day, which will allow their muscles to adjust to the electrical stimulation and help prevent fatigue. During the remaining eight weeks participants will be instructed to use the system all day, when walking at home and in the community.

Participants will have their walking speed and heart rate measured during a 10-metre straight line walking test and a 4-minute figure-8 walking test at baseline, weeks 4, 8 and 12. Participants will perform both tests at each time point without and with the L300 Foot Drop System. Participant satisfaction will be assessed at the end of the 12-week trial.

ELIGIBILITY:
Inclusion Criteria:

* Have multiple sclerosis for at least one year
* Being 18 years of age or older
* Have upper motor neuron-type foot drop (based on the study clinician's medical opinion)
* Able to ambulate at least 10 metres independently or with one person assistance, with or without walking aid
* Having the cognitive capacity to understand and follow the study protocol

Exclusion Criteria:

* Severe cardio-respiratory difficulties (including using a pace-maker) or other health issues that may prohibit walking training
* Significant lower motor neuron neuropathy (based on the study clinician's medical opinion)
* History of frequent falls (more than once a week)
* Having used functional electrical stimulation to treat gait within the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Speed during the 10-metre straight line walking test | 12 weeks
  During the 10-metre straight line walking test, participants walk 10 metres, as marked on the floor with tape, at a steady, self-selected pace, with room for acceleration and deceleration before and after the test. The test measures walking speed, which assesses overall gait function and stability. Participants will complete this test both with and without using the L300 device.

SECONDARY OUTCOMES:
Distance travelled during the 4-minute figure-8 walking test | 12 weeks
  During the 4-minute figure-8 walking test, participants walk at a self-selected speed around a figure-8 track as many times as they can during the four-minute test. The test measures speed, balance, stability and coordination, since it incorporates turning.
Speed during the 10-metre straight line walking test | 4 weeks
  During the 10-metre straight line walking test, participants walk 10 metres, as marked on the floor with tape, at a steady, self-selected pace, with room for acceleration and deceleration before and after the test. The test measures walking speed, which assesses overall gait function and stability. Participants will complete this test both with and without using the L300 device. This timepoint will assess the initial effects of the L300 device.
Speed during the 10-metre straight line walking test | 8 weeks
  During the 10-metre straight line walking test, participants walk 10 metres, as marked on the floor with tape, at a steady, self-selected pace, with room for acceleration and deceleration before and after the test. The test measures walking speed, which assesses overall gait function and stability. Participants will complete this test both with and without using the L300 device.
Distance travelled during the 4-minute figure-8 walking test | 4 weeks
  During the 4-minute figure-8 walking test, participants walk at a self-selected speed around a figure-8 track as many times as they can during the four-minute test. The test measures speed, balance, stability and coordination, since it incorporates turning. This timepoint will assess the initial effects of the L300 device.
Distance travelled during the 4-minute figure-8 walking test | 8 weeks
  During the 4-minute figure-8 walking test, participants walk at a self-selected speed around a figure-8 track as many times as they can during the four-minute test. The test measures speed, balance, stability and coordination, since it incorporates turning.
Physiological cost index during walking tests | 4 weeks
  Based on heart rate, this will assess the physiological cost of walking, as compared to baseline.
Physiological cost index during walking tests | 8 weeks
  Based on heart rate, this will assess the physiological cost of walking, as compared to baseline.
Physiological cost index during walking tests | 12 weeks
  Based on heart rate, this will assess the physiological cost of walking, as compared to baseline.
Participant satisfaction questionnaire score | 12 weeks
  The satisfaction questionnaire will assess participant satisfaction with the L300 Foot Drop System. It will include information about ease of use and desire to continue using the system.
Treadmill Gait Assessment | 12 weeks
  Participants will walk on a standard treadmill at a slow, comfortable speed between 0.5 to 0.8 m/s for one minute. The treadmill is instrumented with an unobtrusive pressure mapping system (Vista Medical Ltd) under the treadmill belt. The pressure mapping system records the centre of foot pressure for each step, which is used to compute step length and width, step time and swing time for 30 consecutive steps. These spatio-temporal gait variables are used to quantify gait performance. This assessment will be completed at baseline and week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Karen D Ethans, MD, Principal Investigator — Health Sciences Centre, Winnipeg; Jessie R Shea, MSc, Study Director — Health Sciences Centre, Winnipeg
Locations (1):
- Rehabilitation Hospital, Health Sciences Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Laufer Y, Hausdorff JM, Ring H. Effects of a foot drop neuroprosthesis on functional abilities, social participation, and gait velocity. Am J Phys Med Rehabil. 2009 Jan;88(1):14-20. doi: 10.1097/PHM.0b013e3181911246. PMID 19096288
- [Background] Ring H, Treger I, Gruendlinger L, Hausdorff JM. Neuroprosthesis for footdrop compared with an ankle-foot orthosis: effects on postural control during walking. J Stroke Cerebrovasc Dis. 2009 Jan;18(1):41-7. doi: 10.1016/j.jstrokecerebrovasdis.2008.08.006. PMID 19110144
- [Background] Stein RB, Everaert DG, Thompson AK, Chong SL, Whittaker M, Robertson J, Kuether G. Long-term therapeutic and orthotic effects of a foot drop stimulator on walking performance in progressive and nonprogressive neurological disorders. Neurorehabil Neural Repair. 2010 Feb;24(2):152-67. doi: 10.1177/1545968309347681. Epub 2009 Oct 21. PMID 19846759
- [Background] O'Dell MW, Dunning K, Kluding P, Wu SS, Feld J, Ginosian J, McBride K. Response and prediction of improvement in gait speed from functional electrical stimulation in persons with poststroke drop foot. PM R. 2014 Jul;6(7):587-601; quiz 601. doi: 10.1016/j.pmrj.2014.01.001. Epub 2014 Jan 9. PMID 24412265